CLINICAL TRIAL: NCT06150339
Title: The OASIS Walking Study - Older Adults With Cognitive Impairment Performing Sit to Stands and Walking in Transitional Care Programs: A Feasibility Study
Brief Title: Older Adults With Cognitive Impairment Doing Sit to Stands, Walking in Transitional Care Programs: A Feasibility Study
Acronym: OASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-5543
Record Dates: First submitted 2023-10-27; First posted 2023-11-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Impairment; Dementia; Delirium; Functional Decline
Keywords: Cognitive Impairment; Dementia; Delirium; Functional Decline; Walking; Walking Program; Activity; Sit to Stand; Chair Stand; Nurse-led; Mobility; Feasibility; Intervention; Quasi-experimental
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Delirium; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a feasibility study which will use a quasi-experimental one group time series design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term Care Stream or Rehab Stream Intervention Arm (Experimental): Intervention Dose: Up to 45 minutes per session, 5 sessions per week, for 6 weeks. Approximately up to 30 minutes will be spent walking; up to 15 minutes will be spent performing sit-to-stands.
  Intervention Components:
  Component 1: Patient-Centered Communication Care Plan. A patient-centered communication care plan will be created, to promote enjoyment and engagement during the sessions. The care plan will be informed by interviews with the participant and their care partner.
  Component 2: Sit to Stand Activity. A target number of sit to stands per session will be determined based on a baseline assessment and according to an algorithm; the target will be progressed halfway into the intervention.
  Component 3: Walking Program. Based on the findings from the patient-centered assessment interviews as well as the performance of the participants on a walk test at baseline (Time 1), an individualized walking program will be carried out with participants.
  Interventions: Other: OASIS Walking Intervention
- Reactivation Stream Intervention Arm (Experimental): Intervention Dose: up to 45 minutes per session, five sessions per week, for 3 weeks. Approximately up to 30 minutes will be spent walking with the participant and up to 15 minutes will be spent performing the sit-to-stands.
  Component 1: Patient-Centered Communication Care Plan. A patient-centered communication care plan will be created, to promote enjoyment and engagement during the sessions. The care plan will be informed by interviews with the participant and their care partner.
  Component 2: Sit to Stand Activity. A target number of sit to stands per session will be determined based on a baseline assessment and according to an algorithm; the target will be progressed halfway into the intervention.
  Component 3: Walking Program. Based on the findings from the patient-centered assessment interviews as well as the performance of the participants on a walk test at baseline (Time 1), an individualized walking program will be carried out with participants.
  Interventions: Other: OASIS Walking Intervention

INTERVENTIONS:
Other: OASIS Walking Intervention — Communication Care Plan, Sit to Stand Activity, Walking Program

SUMMARY:
The goal of this intervention study is to test the effects of a nurse-led mobility intervention (known as the OASIS Walking Intervention (Older Adults performing Sit to Stands and Walking Intervention)) in older adults with cognitive impairment, such as dementia, in transitional care programs.

The main questions this study aims to answer are:

* Is the study doable and are older adults satisfied with the intervention?
* Does the intervention improve older adults' muscle strength, mobility, functional status and quality of life?

Participants will be asked to do the following:

1. Be interviewed once so that a patient-centred communication care plan can be made
2. Do sit to stand activity
3. Walk as part of a walking program.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of and satisfaction of participants with a novel intervention - the OASIS Walking Intervention (that is, the Older Adults with cognitive impairment performing Sit to Stands and Walking Intervention) in a facility-based TCPs.

The second aim is to determine the efficacy of the OASIS Walking intervention on muscle strength, mobility, functional status, quality of life, and discharge destination.

A feasibility study will be undertaken for this three-component intervention project. In terms of study design, a quasi-experimental one group time series design will be used.

A sample size of 26 patient participants and their substitute decision makers will participate in the study. Participants will be older adults ≥65 years admitted to a facility-based transitional care unit in Ontario.

The Older Adults with cognitive impairment performing the Sit to Stands and Walking Intervention is a nurse-led intervention that consists of three components: 1) Patient-Centered Communication Care Plan (informed by interviews with the participant and their care partner); 2) Sit to Stand Activity; and 3) Walking program. This intervention is grounded using a patient centered approach.

For patients in the Long-Term Care Stream or Rehab Stream Arm, the dose of the intervention is: up to 45 minutes per session, five sessions per week, for six weeks. Approximately up to 30 minutes will be spent walking with the participant and up to 15 minutes will be spent performing the sit-to-stand activity.

For patients in the Reactivation Stream Intervention Arm, the dose of the intervention is: up to 45 minutes per session, five sessions per week, for three weeks. Approximately up to 30 minutes will be spent walking with the participant and up to 15 minutes will be spent performing the sit-to-stand activity.

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 years and older;
2. have cognitive impairment (dementia, delirium, cognitive impairment, or unspecified cognitive impairment) as documented in the medical record or Quick Dementia Rating Scale (QDRS) score of ≥2)
3. admitted to a transitional care unit after a hospitalization
4. can speak English
5. has received clearance from the physiotherapist to participate in the study
6. has received clearance from the nurse practitioner to participate in the study
7. were community-dwelling (lived in a home or retirement home; not a nursing home) prior to hospitalization
8. were able to walk independently or with the assistance of one person (with or without a gait aid) prior to hospital admission
9. is currently able to ambulate either independently or with the assistance of one person (with or without a gait aid)
10. has a care partner (family member, friend) who is willing participate in an interview about the patient for the study.

Exclusion Criteria:

1) Palliative (having <six months prognosis as documented in the medical chart)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From start of recruitment to end of recruitment (6 months)
  Recruitment rate will be calculated as the percentage of participants who enroll in the study out of the total number of eligible participants
Retention rate | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  Retention rate will be calculated as the percentage of participants who complete the study (i.e., receive the full dose of the intervention and provided post-test outcome data) out of the number of participants who were enrolled (i.e., signed a consent form and provided baseline data)
Adherence (Level of engagement with the treatment [percentage]). | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  The level of engagement with the treatment (percentage). For this study, the planned number of sessions is five per week for 6 weeks for a total of 30 sessions.
  Percentage = the number of sessions attended divided by the total number of sessions (30 sessions)
Adherence (Average number of treatment sessions attended) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  Average number of treatment sessions attended
Adherence (Average duration of each intervention session) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  The average duration of each intervention session (in minutes)
Adherence (Average duration of each walking session) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  The average duration of each walking session (in minutes)
Adherence (Average number of sit to stands done per session) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  Average number of sit to stands done per session.
Adherence (Level of engagement with sit to stands [percentage]) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  Percentage = number of sit to stands done per session, divided by the goal number of sit to stands.

SECONDARY OUTCOMES:
Participant Satisfaction (for Long-Term Care Stream or Rehab Stream Arm) | Posttest (Immediately after 6-week intervention) (Time 3)
  8-Item Client Satisfaction Questionnaire (CSQ-8) + 3 Open-Ended Questions. The CSQ-8 has a minimum value is 8, the maximum value is 32. Higher scores mean a better outcome.
Participant Satisfaction (for Reactivation Stream Intervention Arm) | Posttest (Immediately after 3-week intervention) (Time 3)
  8-Item Client Satisfaction Questionnaire (CSQ-8) + 3 Open-Ended Questions. The CSQ-8 has a minimum value is 8, the maximum value is 32. Higher scores mean a better outcome.
Lower extremity muscle strength (for Long-Term Care Stream or Rehab Stream Arm) | Pretest Initial Assessment (Time 1); After 3 weeks of intervention (Time 2); Posttest (Immediately after 6-week intervention) (Time 3)
  time to perform one sit-to-stand
Lower extremity muscle strength (for Reactivation Stream Intervention Arm) | Pretest Initial Assessment (Time 1); After 1.5 weeks of intervention (Time 2); Posttest (Immediately after 3-week intervention) (Time 3)
  time to perform one sit-to-stand
Mobility (for Long-Term Care Stream or Rehab Stream Arm) | Pretest Initial Assessment (Time 1); After 3 weeks of intervention (Time 2); Posttest (Immediately after 6-week intervention) (Time 3)
  2-minute walk test
Mobility (for Reactivation Stream Intervention Arm) | Pretest Initial Assessment (Time 1); After 1.5 weeks of intervention (Time 2); Posttest (Immediately after 3-week intervention) (Time 3)
  2-minute walk test
Functional Status (for Long-Term Care Stream or Rehab Stream Arm) | Pretest Initial Assessment (Time 1); After 3 weeks of intervention (Time 2); Posttest (Immediately after 6-week intervention) (Time 3)
  Barthel Index (BI). The BI has a minimum value of 0 and a maximum value of 20. Higher scores mean a better outcome.
Functional Status (for Reactivation Stream Intervention Arm) | Pretest Initial Assessment (Time 1); After 1.5 weeks of intervention (Time 2); Posttest (Immediately after 3-week intervention) (Time 3)
  Barthel Index (BI). The BI has a minimum value of 0 and a maximum value of 20. Higher scores mean a better outcome.
Patient's Quality of Life (for Long-Term Care Stream or Rehab Stream Arm) | Pretest Initial Assessment (Time 1); After 3 weeks of intervention (Time 2); Posttest (Immediately after 6-week intervention) (Time 3)
  The Quality of Life-AD Measure (QOL-AD). The QOL-AD is a 13-item questionnaire. Participants rate each item on a 4-point scale, with 1 being poor and 4 being excellent. The minimum score is 13 and the maximum score is 52. Higher scores mean a better outcome.
Discharge destination (for Long-Term Care Stream or Rehab Stream Arm) | At the time of discharge from the TCU or within 60 days of admission to TCP, whichever comes first.
  Discharge destination after TCP
Discharge destination (for Reactivation Stream Intervention Arm) | At the time of discharge from the TCU or within 60 days of admission to TCP, whichever comes first.
  Discharge destination after TCP
Intervention fidelity (percentage) | Calculated at the end of the study (6 months + 6 weeks from the start of recruitment)
  Intervention fidelity will also be measured through the interventionist's self-report of 12 intervention items. The percentage will be calculated as the number of items done divided by the 12 items on the intervention fidelity checklist. Minimum value is 0%, maximum value is 100%. A higher percentage means a better outcome (greater intervention fidelity).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S McGilton, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Abbeylawn Retirement Home Transitional Care Unit (Operated by Bayshore Health Care), Pickering, Ontario
  - Cedarbrook Lodge Retirement Home Transitional Care Unit (Operated by Bayshore Health Care), Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cumal A, Colella TJF, Puts MT, McGilton KS. The OASIS walking study-Older adults with cognitive impairment performing sit to stands and walking in transitional care programs: Protocol for a feasibility study. PLoS One. 2024 Sep 16;19(9):e0308268. doi: 10.1371/journal.pone.0308268. eCollection 2024. PMID 39283901